CLINICAL TRIAL: NCT07378826
Title: Comparison of Power Training Progression Methods in Older Independently Living Adults.
Brief Title: Power Training Progression Methods
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Joseph Signorile, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20251334
Record Dates: First submitted 2026-01-22; First posted 2026-01-30 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Activity, Motor
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RPE-Based Power Training (Active Comparator): The RPE system will be based on movement speed with an unloaded condition producing maximal speed (RPE=10) and a 1RM producing minimal speed (RPE = 1). If RPE is above 5, loads will be increased by 5% for upper body exercises and 2.5% for lower body exercises. If the RPE = between 4 and 5 the load will remain unchanged. If RPE falls below 4, loads will be lowered using the same percentages.
  Interventions: Behavioral: RPE-Based Power Training
- Power Plateau-Based Power Training (Active Comparator): Following two training sessions, the average power for each exercise will be calculated. When average power increases by a minimum of 5% from session one to session two, the load will remain unchanged to continue to reap power improvements. When the average power does not increase by at least 5% from session one to two, the load will be increased by the same protocol described above. Loads will only decrease when subjects cannot complete all repetitions with adequate form.
  Interventions: Behavioral: Power Plateau-Based Power Training

INTERVENTIONS:
Behavioral: RPE-Based Power Training — The RPE system will be based on movement speed with an unloaded condition producing maximal speed (RPE=10) and a 1RM producing minimal speed (RPE = 1). If RPE is above 5, loads will be increased by 5% for upper body exercises and 2.5% for lower body exercises. If the RPE = between 4 and 5 the load will remain unchanged. If RPE falls below 4, loads will be lowered using the same percentages.
  Arms: RPE-Based Power Training
Behavioral: Power Plateau-Based Power Training — Following two training sessions, the average power for each exercise will be calculated. When average power increases by a minimum of 5% from session one to session two, the load will remain unchanged to continue to reap power improvements. When the average power does not increase by at least 5% from session one to two, the load will be increased by the same protocol described above. Loads will only decrease when subjects cannot complete all repetitions with adequate form.
  Arms: Power Plateau-Based Power Training

SUMMARY:
This study will investigate the impact of two unique progression models for power training in a sample of healthy older adults. The objective is to identify the most practical methodology for implementing power training, which is considered a critical marker of functional capacity in older populations.

ELIGIBILITY:
Inclusion Criteria:

* 50 - 90 years of age.
* Be able to walk 50m without any sort of assistance device.
* Be able to understand and communicate in English to properly conduct the training and testing processes.

Exclusion Criteria:

* Uncontrolled cardiovascular or neuromuscular disease that prevent participation in a training program.
* Any systemic inflammatory or autoimmune conditions such as rheumatoid arthritis, or other serious concomitant medical illness.
* Unresolved injury or surgery to the upper or lower limbs that prevents weight training.
* - Montreal Cognitive Assessment (MoCA) score below 18

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2026-01-30 (Actual); Primary Completion 2027-05-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Change in neuromuscular performance as measured by 1-repetition maximum (1RM) | Baseline, 12 weeks
  Maximal load that can be lifted in one repetition (1RM) will be assessed in both leg press and chest press exercises. The loads on the testing equipment will be increased across 5 to 7 testing repetitions. The persons 1RM will be the highest load the person can move through the range of motion of the exercise. There are no minimum or maximum scores for this test. The higher the 1RM the stronger the person is. The unit of measurement is kilograms.
Change in neuromuscular performance as measured by Watts | Baseline, 12 weeks
  This test measures the power a person can produce at maximal speed using loads of 20%, 40%, 60%, 80%, and 90% of 1RM for the chest press and leg press. Power shows how fast a person can do work. Unit of measure is Watts.

SECONDARY OUTCOMES:
Change in the Speed of the Ten-Meter Walk Test. | Baseline, 12 weeks
  The ten-meter walk test will be used to assess gait velocity. The participants will be asked to walk at usual walking speed and as quickly as possible in a straight line on a 10-m course marked at 0, 2, 8 and 10 m. On verbal command, participants will start on the 0-m mark and stop when the 10-m mark is crossed. The total time to ambulate from the 2-m mark to the 8-m mark (6 m total) will be timed to the hundredth of a second. Two trials will be performed at each speed, and the average will be documented in meters per second. One-minute recoveries will be provided between trials.
Change in Time for the Five Times Sit-to-Stand Test. | Baseline, 12 weeks
  The five-time sit-to-stand test will be used to assess functional lower body strength. The participant will sit with arms folded across the chest and the back against the chair. On a verbal command, the participant will stand up and sit down five times as quickly as possible. Timing begins at the word go and ends when the buttocks touch the chair after the fifth repetition. One practice and two testing trials will be performed. Time will be measured in seconds.
Change in Distance of the Seated Medicine Ball Throw. | Baseline, 12 weeks
  For the Seated Medicine Ball Throw, subjects will sit in an armless chair with the back against the chair back, while holding the 6-pound medicine ball against the chest.
  Subjects will then throw the ball at a perceived 45° angle as far as possible. Subjects must complete at least three practice trials; however, subjects will be allowed more trials until comfortable with the testing procedure. Upon starting the official trial, subjects will complete three separate attempts at each varying medicine ball, to nine trials in total.
  Each of the three trials within a given medicine ball test will be separated by a 1-minute rest. Distance will be measured in centimeters
Change in the time required to complete the timed Up-and-Go Test. | Baseline, 12 weeks
  Upon verbal cue, the subject stands up, walks around a cone placed three meters from the front edge of the chair and then returns to a seated position as quickly as possible. Time is measured in seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph F. Signorile, PhD, Principal Investigator — University of Miami
Locations (1):
- Laboratory of Neruomuscular Research and Active Aging, Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: No